CLINICAL TRIAL: NCT03122548
Title: A Phase 2, Open-label Evaluation of CRS-207 and Pembrolizumab in Adults With Recurrent or Metastatic Gastric, Gastroesophageal Junction, or Esophageal Adenocarcinomas
Brief Title: Safety and Efficacy of CRS-207 With Pembrolizumab in Gastric, Gastroesophageal Junction or Esophageal Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment and lack of clinical activity in other CRS-207 studies.
Sponsor: Aduro Biotech, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-14; KEYNOTE KN-463 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2017-04-04; First posted 2017-04-21 (Actual); Results first posted 2019-02-20 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: stomach cancer; gastric cancer; esophageal cancer; digestive system diseases; gastrointestinal diseases; stomach diseases
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms; Esophageal Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Stomach Diseases | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CRS-207 + Pembrolizumab (Experimental): CRS-207 and pembrolizumab will be administered in 3-week cycles. For Cycle 1, pembrolizumab (200 mg) will be administered by intravenous (IV) infusion over 30 minutes on Day 1 and CRS-207 (starting dose 1 × 10e9 colony-forming units [CFU]) will be administered by IV infusion over 1 hour on Day 2. If the infusions are well tolerated, pembrolizumab and CRS-207 may be administered on the same day (Day 1) for subsequent cycles. After 4 cycles, pembrolizumab will continue to be administered on Day 1 at each treatment cycle (every 3 weeks); CRS-207 will be administered once every 6 weeks (every other cycle). Treatment will continue for up to 35 cycles as long as there is adequate safety and potential for clinical benefit.
  Interventions: Biological: CRS-207; Biological: Pembrolizumab

INTERVENTIONS:
Biological: CRS-207 — Administered by IV infusion over 1 hour.
Biological: Pembrolizumab — Administered by IV infusion over 30 minutes.
  Other Names: MK-3475

SUMMARY:
The purpose of this study is to determine whether CRS-207 in combination with pembrolizumab is safe and effective in adults with recurrent or metastatic gastric, gastroesophageal junction, or esophageal cancer who have received one or two prior chemotherapy regimens for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with confirmed histology of one or more of the following:

   * Histologically-confirmed gastric or gastroesophageal junction (GEJ) adenocarcinoma (Siewert type II/III classification), or
   * Histologically-confirmed inoperable superior, medial, or distal third esophageal adenocarcinoma (Siewert type I classification may be included, provided there is no mixed histology)
2. Confirmed recurrent or metastatic disease
3. Received and experienced disease progression on, or following one or two prior chemotherapy regimens for advanced disease.
4. HER-2/neu negative or, if HER-2/neu positive, disease must have previously progressed on treatment with trastuzumab; prior treatment must have included a platinum and a fluoropyrimidine.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Can provide tissue for PD-L1 and mesothelin biomarker analysis
7. Adequate organ and marrow function at screening

Exclusion Criteria:

1. Diagnosis of squamous or undifferentiated gastric cancer
2. Individuals with inaccessible tumors or for whom biopsy is contraindicated
3. Participated in any other study in which receipt of an investigational new drug or investigational device occurred within 28 days of first dose of study drug
4. Receiving tumor necrosis factor (TNF) pathway inhibitors, PI3 kinase inhibitors, systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
5. Clinical evidence of ascites by physical exam
6. Prior anti-cancer monoclonal antibody within 4 weeks prior to first dose of study drug or has not recovered from adverse effects due to agents administered more than 4 weeks earlier
7. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to first dose of study drug, or has not recovered from adverse effects due to a previously-administered agent
8. Subjects who have implanted medical devices that pose high risks for colonization and cannot be easily removed (e.g. artificial heart valves, pacemakers, prosthetic joints, orthopedic screw(s), metal plate(s)) if infection occurs. Other common devices such as venous access devices (e.g. Port-a-Cath or Mediport) may be permitted as well as arterial and venous stents and dental and breast implants that were placed more than 3 months prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mary Crowley Cancer Research, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CRS-207 + Pembrolizumab: Treatment cycle is once every 3 weeks. Pembrolizumab: 200 mg administered by intravenous (IV) infusion on Day 1 of each 3-week cycle. CRS-207: 1×10e9 colony forming units (CFU) administered by IV infusion on Day 2 of Cycle 1, Day 1 of Cycles 2, 3, 4, and Day 1 every 6 weeks thereafter (every other cycle).
Period: Overall Study
Arm/Group | CRS-207 + Pembrolizumab
Started | 5
Completed | 0
Not Completed | 5
Not completed — Death | 2
Not completed — Progression - subject went into hospice | 1
Not completed — Study Terminated by Sponsor | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics provided for all subjects who were administered at least 1 dose of protocol-specified drug (the Safety Analysis Set [SAF]).
Groups:
- CRS-207 + Pembrolizumab: Treatment cycle is once every 3 weeks. Pembrolizumab: 200 mg administered by IV infusion on Day 1 of each 3-week cycle. CRS-207: 1×10e9 CFU administered by IV infusion on Day 2 of Cycle 1, Day 1 of Cycles 2, 3, 4, and Day 1 every 6 weeks thereafter (every other cycle).
Arm/Group | CRS-207 + Pembrolizumab
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was evaluated based upon the best overall response (BOR) for individual study subjects. BOR was determined by the highest post-baseline qualitative response value for each evaluable subject as measured by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) and given the following hierarchy of overall response results: complete response (CR) > partial response (PR) > stable disease (SD) > progressive disease (PD) > not evaluable (NE). The protocol-specified ORR was defined as the percentage of evaluable subjects with a BOR of CR or PR; however, this percentage was not calculated per the final study Statistical Analysis Plan (SAP). Therefore, the number of evaluable subjects with BOR RECIST v1.1 values of CR, PR, SD, PD, and NE are provided for this outcome measure. .
Time Frame: BOR was assessed from the first post-baseline tumor assessment until documented disease progression, starting of a new cancer treatment, death, or study termination, whichever is earlier, assessed up to 15 weeks.
Population: Analysis based upon subjects who received at least 1 dose of CRS-207 and had at least 1 evaluable post-baseline RECIST v1.1 tumor response assessment or were discontinued due to toxicity (the Evaluable Analysis Set [EAS]). 2 subjects did not have post-baseline tumor response assessments and could not be evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CRS-207 + Pembrolizumab
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0
  Progressive Disease | 3
  Not Evaluable | 0

2. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of evaluable subjects who exhibited a post-baseline tumor assessment BOR rating of CR, PR, or SD per RECIST v1.1.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CRS-207 + Pembrolizumab
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Number of weeks from the date of first dose of study treatment to the first date of objectively determined progressive disease (PD) according to RECIST v1.1 or death from any cause, estimated using Kaplan-Meier (KM) methods with 95% confidence intervals (CIs). Subjects who do not experience PD and are alive on or before the data cut-off date will be censored at the time of last evaluable tumor assessment or data cut-off date, whichever is earlier.
Time Frame: Subjects followed for disease progression from first dose of study treatment until documented disease progression, initiation of new cancer treatment, death, or study termination, whichever is earlier, assessed up to 15 weeks.
Population: Analysis of PFS was performed on subjects in the SAF.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CRS-207 + Pembrolizumab
Number analyzed (Participants) | 5
weeks | 5.43 [0.14 to 6.00]

4. Secondary Outcome: Duration of Response (DOR)
Description: Number of weeks from the first date a study subject achieved an objective disease response of CR or PR according to RECIST v1.1 to the date a study subject exhibited PD or death due to any cause, estimated using KM methods with 95% CIs. Subjects who do not experience PD or death at the time of analysis will be censored at the time of last evaluable tumor assessment or data cut-off date, whichever is earlier.
Time Frame: DOR assessed from the date of a post-baseline tumor assessment of CR or PR per RECIST v1.1 until the date of documented disease progression, starting of a new cancer treatment, death, or study termination, whichever is earlier, assessed up to 15 weeks.
Population: No study subjects achieved CR or PR designation, therefore, per the final SAP DOR was not derived.
Measure: Count of Participants; unit: Participants
Arm/Group | CRS-207 + Pembrolizumab
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Number of weeks from the date of first dose of study treatment to the date of death from any cause, estimated using KM methods with 95% CIs for subjects in the SAF. Subjects without documentation of death at the time of analysis were censored as of the date the subject was last known to be alive, or the data cut-off date, whichever is earlier.
Time Frame: OS was assessed from the first dose of study treatment until death or study termination, whichever is earlier, assessed up to 15 weeks.
Population: Analysis of OS was performed on subjects in the SAF.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CRS-207 + Pembrolizumab
Number analyzed (Participants) | 5
weeks | 11.57 [4.00 to 14.43]

ADVERSE EVENTS:
Time Frame: Subjects were followed for serious and non-serious adverse events (AEs) from the beginning of any study treatment until 28 days following the last dose of study drug or until the subject initiates a new cancer therapy, whichever is earlier, an average of 3 months. Subjects were followed for survival for at least 12 months after end-of-treatment (EOT), or until death, loss to follow-up, or study termination, whichever is earlier, an average of 10 weeks.
Description: AEs reported for the SAF. Methods of determining whether certain AEs have occurred include regular investigator assessment and regular laboratory testing.
Arm/Group | CRS-207 + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CRS-207 + Pembrolizumab (N=5)
Obstruction Gastric (Gastrointestinal disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Hepatic Encephalopathy (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CRS-207 + Pembrolizumab (N=5)
Chills (General disorders) | 4
Pyrexia (General disorders) | 4
Fatigue (General disorders) | 3
Oedema Peripheral (General disorders) | 2
Pain (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Obstruction Gastric (Gastrointestinal disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hepatic Encephalopathy (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1
Blood Sodium Decreased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 1
Weight Decreased (Investigations) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated early and included a small number of subjects, and insufficient data were available to evaluate the clinical activity of the study treatment. Due to low enrollment, some protocol-specified outcome measures were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction is that study results will first be published in a joint multi-center paper unless (a) written confirmation is provided to the site or PI indicating that there will be no multi-center publication, or (b) at least 12 months have passed after the completion of data analysis at all study sites. Publications will be submitted for sponsor review ≥ 30 days prior to the publication date. Sponsor cannot require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT03122548/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03122548/SAP_001.pdf